CLINICAL TRIAL: NCT04511884
Title: Screening Microorganism of Cryptogenic Mechanical Pneumonia Through NGS to Lung Tissue Fluid
Brief Title: Screening Microorganism of Cryptogenic Mechanical Pneumonia Through Next Generation Sequencing to Lung Tissue Fluid
Acronym: COPandNGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director of respiratory and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2020040695
Record Dates: First submitted 2020-04-26; First posted 2020-08-13 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cryptogenic Organizing Pneumonia; Idiopathic Interstitial Pneumonias
Keywords: cryptogenic organizing pneumonia; next-generation sequencing
MeSH Terms: conditions — Cryptogenic Organizing Pneumonia; Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing — The patient who may be diagnosed with cryptogenic organizing pneumonia will be detected through next-generation sequencing.

SUMMARY:
The etiology of cryptogenic organizing pneumonia (COP)was not clear, but previous studies have shown that in some patients, some pathogen could be detected in bronchoalveolar lavage fluid (BALF), and may be one of the causes of COP. This study aimed to screen the pathogenic microorganisms in BALF and lung puncture fluid of the patients with COP through the next-generation sequencing to further clarify the correlation between the incidence of COP and pathogenic microorganisms.

DETAILED DESCRIPTION:
The cause of cryptogenic organizing pneumonia (COP) was unknown, but studies had shown that certain bacteria, viruses, or specific pathogens could be detected in bronchoalveolar lavage fluid (BALF) in some patients, and these pathogenic microorganisms may be the cause of COP. Specimens were obtained by conventional methods (sputum, blood, BALF or lung puncture fluid) for microbiological detection. Due to the influence of the quality of acquired specimens, specimen preservation and transportation which were influenced by external factors, many patients did not get good test results, which affected the diagnosis and subsequent treatment of patients. Next-generation sequencing (NGS) which could determine hundreds of thousands to millions of DNA molecules in parallel at one time, and efficiently sequence or fragment of pathogenic microorganisms. NGS had greatly improved the detection rate of pathogenic microorganisms. This study aimed to screen pathogenic microorganisms in BALF and lung puncture fluid of COP patients by NGS, and further clarify the correlation between occurrence of COP and pathogenic microorganisms.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was older than 18 years old.
2. The patient was organizing pneumonia (OP) through pathology.
3. The patient was diagnosed as OP from clear cause through routine detection.
4. Chest CT shows consolidation or ground glass

Exclusion Criteria:

1. The patient has specific characteristics of connective tissue disease or autoimmune disease.
2. The patient has a clear other cause of OP.
3. The patient has severe systemic diseases of heart, brain, liver, kidney and so on, and cannot tolerate invasive examination
4. The patient disapproves of invasive testing

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with cryptogenic organizing pneumonia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of microorganisms positive for cryptogenic organizing pneumonia detected by NGS | From 1 Dec 2019 to 1 Dec 2024
  The patients with cryptogenic organizing pneumonia will be detected through electronic bronchoscopy and lung puncture. The sample will be examinated through NGS.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - BAI Jiu-wu, Shanghai, Please Select
  - Shanghai Pulmonary Hospital, Tongji University, Shanghai, Shanghai Municipality